CLINICAL TRIAL: NCT06520826
Title: Safety of Three Times Weekly Oral Vadadustat for the Treatment of Anemia in Hemodialysis Subjects: Vafseo Outcomes In-Center Experience
Brief Title: Vafseo Outcomes In-Center Experience
Acronym: VOICE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: USRC Kidney Research (Network)
Collaborators: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USRC-2024-001
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Anemia of Chronic Kidney Disease
MeSH Terms: interventions — vadadustat; Hematinics; Epoetin Alfa; continuous erythropoietin receptor activator; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vadadustat (Experimental): Vadadustat, 300 mg tablets, administered orally three times per week
  Interventions: Drug: Vadadustat
- Erythropoiesis-stimulating agent (ESA) - Standard of Care (SOC) (Active Comparator): Epoetin alfa (EPOGEN), Methoxy polyethylene glycol-epoetin beta (Mircera), or Darbepoetin alfa (Aranesp) administered as per standard of care
  Interventions: Drug: Erythropoiesis Stimulating Agent

INTERVENTIONS:
Drug: Vadadustat — A synthetic, orally bioavailable, small molecule being developed as an inhibitor of hypoxia-inducible factor prolyl-hydroxylases for the treatment of anemia associated with chronic kidney disease. Intervention to be administered to maintain hemoglobin within a target range of 10-11 g/dL.
  Other Names: Vafseo
  Arms: Vadadustat
Drug: Erythropoiesis Stimulating Agent — Standard of care erythropoiesis stimulating agent will be administered to maintain hemoglobin within a target range of 10-11 g/dL.
  Other Names: Epoetin alfa (EPOGEN), Methoxy polyethylene glycol-epoetin beta (Mircera), or Darbepoetin alfa (Aranesp)
  Arms: Erythropoiesis-stimulating agent (ESA) - Standard of Care (SOC)

SUMMARY:
This trial is an investigator-initiated, multi-center, randomized (1:1), open-label, active-controlled, pragmatic study of the safety of vadadustat administered three times per week for the treatment of anemia in in-center hemodialysis patients with End Stage Kidney Disease (ESKD). This study will obtain long-term safety data in a large sample of subjects receiving in-center hemodialysis to support adoption of three times per week vadadustat dosing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than or equal to 18 years of age.
* Receiving outpatient in-center hemodialysis at least three times per week for end-stage kidney disease.
* Currently prescribed or eligible for erythropoiesis-stimulating agent based on approved facility policy
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

* Contraindication to receive vadadustat or any of its known constituents per USPI.
* Cirrhosis or active, acute liver disease. Concomitant use of any hypoxia-inducible factor prolyl-hydroxylases or OAT1/OAT3 inhibitors (probenacid, rifampicin, gemfibrozil, or teriflunomide).
* Unable to comply with study requirements or in the opinion of a healthcare provider or a member of the central study team, not clinically stable to participate in the study.
* Pregnant at time of consent (per subject self-report).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 18 months

SECONDARY OUTCOMES:
All-cause hospitalization | 18 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - USRC Kidney Research, Lone Tree, Colorado
  - Nephrology and Hypertension Specialists, PC, Dalton, Georgia
  - US Renal Care - Gallup, Gallup, New Mexico
  - Dallas Renal Group, Dallas, Texas
  - US Renal Care - Live Oak, Live Oak, Texas